CLINICAL TRIAL: NCT04043689
Title: Therapeutic Effects of Transcranial Alternative Current Stimulation (tACS) in Chronic Post Stroke Hemianopia
Acronym: HEMIANOTACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP 190051; 2019-A00501-56 (Other: N°IDRCB)
Record Dates: First submitted 2019-07-25; First posted 2019-08-02 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Hemianopsia
MeSH Terms: conditions — Hemianopsia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- tACS stimulation of the right frontal region (Active Comparator): Active tACS stimulation of the right frontal region (around the right FEF, EEG electrode FC2) at a high-beta frequency (30 Hz) with the goal of visibly training EEG recordings, frontal oscillatory activity and right fronto-parietal synchrony (FEF-IPS, or between FC2 and P4 electrodes) in the high-beta band (~ 30 Hz) which facilitates attentional orientation and visual perception in the two visual hemi-fields, but more particularly the targets present on the blind field of vision.
  Interventions: Device: tACS (transcranial Alternate Current Stimulation)
- tACS stimulation of the occipito-parietal region (Active Comparator): Active tACS stimulation of the occipito-parietal posterior contralesional region(around the right IPS, EEG electrode P4), at an alpha frequency (10 Hz) which will induce on the EEG recordings an oscillatory drive in the alpha band ( ~ 10Hz) and an increase in synchrony at this frequency band on the stimulated posterior occipital and parietal lobe (EEG electrodes P4 and 02), but also, by transcallosal push-and-pull phenomena, a desynchronization effect of the contralateral posterior occipital and parietal area (EEG electrodes P3 and 01), which will facilitate attention orientation and target detection in the blind visual field of view.
  Interventions: Device: tACS (transcranial Alternate Current Stimulation)
- TACS stimulation of the right frontal (FEF) (Sham Comparator): . Condition TACS stimulation of the right frontal (FEF) at a high-beta frequency (30 Hz) for half of the patients and unilateral occipital cortex (right / left) at an alfa frequency (10 Hz) for the other half . This condition will control the possible placebo effects of tACS stimulation and the potential effects of visual field enhancement with repetition of perimetry tests. This condition will also verify the lack of changes in cerebral rhythm activity in the case of an application without effective electrical current.
  Interventions: Device: tACS (transcranial Alternate Current Stimulation)

INTERVENTIONS:
Device: tACS (transcranial Alternate Current Stimulation) — This is a single-centric comparative randomized controlled blind and cross-over study.
  The order of stimulation conditions will be randomized: (right frontal tACS / occipital tACS / tACS PLACEBO). The 3 stimulation conditions will be performed with a wash-out period of at least 1 week. In this study each patient will be his own control

SUMMARY:
Background: The most common visual field deficit after retro-chiasmatic lesions is homonymous hemianopia (HH), defined as the impossibility of seeing the contralesional visual hemisphere without ocular injury. HH affects between 90000 and 120 000 new cases per year in the United States and Europe HH was reported in 30% of patients after stroke (National Audit Office) (in France, with 130,000 strokes per year, 39,000 patients with HH). Despite the 30-year decline, the rehabilitation techniques have a low level of evidence of their effectiveness and few are used in routine clinical practice in France.

Transcranial Alternate Current Stimulation (tACS) is a method of Alternative Current stimulation that can modulate neural activity by imposing local oscillatory activity.

An observational study of occipital tACS in patients with optic nerve lesions showed an increase in visual field size, power, and occipital alpha synchrony. Two transorbital tACS studies showed visual improvements , and compensations for abnormally weak oscillatory activity by temporal resynchronization. Our team has demonstrated a role of noninvasive brain stimulation in right hemisphere frontal eye fields on cortical beta-high (~ 30 Hz) oscillatory activity, improving the visual perception of both hemi-fields and the fronto-parietal synchrony of the right hemisphere.

Objective:

This project aims to compare, on the same patient population, two tACS stimulation strategies, with the aim of increasing the attentional orientation towards the blind visual hemi-field and thus the visual detection of stimuli in this hemi-field. .

For this, The investigator team will evaluate on the one hand an occipital stimulation (V1-IPS) contralateral to the lesion, at a alfa frequency (10 Hz), which induces the desynchronization of the contralateral hemisphere with the aim of improving the visual perception of targets in the blind visual hemi-field. the study will compare this intervention to a stimulation of the frontal region (FEF) of the right hemisphere at a high-beta frequency (30 Hz), which showed effects of facilitation of endogenous and exogenous attentional orientation. The two previous strategies will be compared to a placebo tACS stimulation session.

DETAILED DESCRIPTION:
Background:

Focusing on low-level perceptual activities, and robust, controlled explorations with medium-sized cohorts, several studies have shown tACS effects related to oscillatory activity and inter-regional synchrony.

For example, in healthy subjects, occipital tACS showed an increase in posterior alpha power following tACS alpha (10-14 Hz). At higher frequencies, the 60 Hz tACS showed a sustained reduction in visual contrast sensitivity threshold . Two studies in 2014 have also shown following 40 Hz tACS stimulation of occipital or parietal brain regions in healthy humans, sustained dependent on synchrony of posterior interhemispheric gamma band networks, and modulation effects of moving target perception Very recently, a 10 Hz occipital tACS stimulation study coupled with functional magnetic resonance Imaging recording (fMRI) showed diffuse effects likely to indicate occipito-parieto-temporal synchronization during the delayed phase of effects.

Among patients' trials, an observational study of uncontrolled occipital tACS in patients with optic nerve lesions showed improved visual acuity and visual field size, accompanied by an increase in power and of occipital alpha synchrony by targeting periorbital regions; More recently, a double-blind, multicenter, controlled trial in patients with optic nerve lesions showed, with daily transorbital tACS sessions lasting 10 weeks, a sustained (2.5%) increase in visual field size versus stimulation placebo.

This project aims to compare, on the same patient population, two tACS stimulation strategies, with the aim of increasing the attentional orientation towards the blind visual hemi-field and thus the visual detection of stimuli in this hemi-field. .

For this, the study will evaluate on the one hand an occipital stimulation (V1-IPS) contralateral to the lesion, at a alfa frequency (10 Hz), which induces the desynchronization of the contralateral hemisphere with the aim of improving the visual perception of targets in the blind visual hemi-field. This intervention will be compared to a stimulation of the frontal region (FEF) of the right hemisphere at a high-beta frequency (30 Hz), which showed effects of facilitation of endogenous and exogenous attentional orientation. The two previous strategies will be compared to a placebo tACS stimulation session.

The overall goal of this project is to modulate visual perception in patients with HH in the chronic phase using transcranial AC stimulation. The study aim is to evaluate the behavioral effects of tACS stimulation of the right fronto-parietal network (FEF-IPS) and the occipital and parieto-occipital region (V1-IPS), contralateral to the lesion, on visual perception in static and kinetic perimetry. The effects of stimulation of these two targets on brain activity by electrophysiology (EEG) will be quantified. The hypothesis is that the tACS, by increasing the functional connectivity (phase synchronism at the frequency delivered during the stimulation), will make it possible to modulate the threshold of visual perception.

Specifically, the hypothesis is that a single session of 30 Hz tACS stimulation of the right frontal cortex (around the right FEF) will increase fronto-parietal synchrony within the right hemisphere of patients with lesions acquired brain responsible for chronic HH, thus improving the static and kinetic visual field in the first 30 minutes post-stimulation. The investigator team also hypothesize that a single session of tACS stimulation on the occipital and posterior parietal cortex contralateral to the lesion (around the V1 region) of patients with acquired brain lesions responsible for chronic HH will improve the visual field in the first 30 minutes post-stimulation, but this improvement will be less compared to the improvement caused by the stimulation of the right FEF, which could be accompanied by a temporary decrease in the visual perception of the targets on the healthy visual hemi-field.

Methods:

Monocentric comparative randomized controlled, cross-over and blinded study, Major population, acquired brain lesion responsible for homonymous hemianopia, chronic phase of cerebrovascular accident (between 3 months and 10 years of evolution) and cohort healthy subjects not treated with tACS to obtain normative data from visual fields, neuroimaging (MRI) and electroencephalography (EEG)

* Each patient or each healthy volunteer will have an inclusion visit including visual static and kinetic perimetry, EEG recordings, cognitive tests, questionnaire and brain MRI.
* Then, each patient will have 3 visits, including a first evaluation period (perimetry, EEG and reading tests) then a stimulation session (right frontal active tACS or contralesional occipito-parietal active tACS, or placebo tACS) then a second evaluation time (EEG, perimetry , and reading tests)

Discussion:

The investigator team expect an immediate and significant increase in visual field size and improved visual detection capabilities of patients treated with active tACS stimulation on the right frontal region (FEF) and / or contralateral occipital region (V1-IPS) lesion

The project will contribute to the development of an innovative treatment to improve the quality of life of HH brain-injured patients, lacking effective treatment options to date.

TACS is an easily accessible and easily applicable technique in large-scale clinical practice. Coupled with EEG monitoring, it is the only one that allows efficient and safe manipulation of oscillatory activity and interregional synchronicity.

Interest in these new methods of non-invasive brain stimulation guiding brain plasticity, in stroke (130,000 new cases / year) or head trauma is very important. The scientific, clinical and technological implications are major.

ELIGIBILITY:
Inclusion Criteria:

Patient aged 18 and over

* Patient with homonymous lateral hemianopia with brain injury acquired for at least 3 months and at most 10 years after ischemic stroke, cerebral hematoma
* Patient able to understand French both orally and in writing
* Patient giving free, informed and written consent
* Absence of a neurological disease interfering with the passing of tests

Non-inclusion criteria :

* Patients subject to a legal protection measure (safeguarding of justice, guardianship and trusteeship, protected adults)
* Pre-existing severe ophthalmological disorders, visual field disorders visual field disorders, monocular visual acuity less than 5/10, severe oculomotor disorders (post-stroke ophthalmological consultation less than at the time of inclusion)
* Contraindication of tACS and / or magnetic resonance imaging (pacemaker or implantable defibrillator, intracranial electrodes or other intracranial implant, cranial vault anomalies facing stimulation electrodes (plates, prostheses, uncovered skull)
* Pregnant women and nursing mothers
* Recruitment in other interventional studies for the duration of the participation.
* Non-affiliation to a social security scheme (excluding AME) or non-beneficiary of such a scheme

Healthy participants inclusion criteria are the following:

* Healthy Subject 18 years and older
* Healthy subject able to understand French both orally and in writing
* Healthy subject who has given free and informed consent and writes

Healthy participants non-inclusion criteria are the following:

* Severe neurological, psychiatric, physical, or ophthalmological disorders (binocular visual acuity less than 5/10, ophthalmological consultation less than one year old at the time of inclusion) that interfere with the normal performance of tests and study tasks
* Contraindication to magnetic resonance imaging (pacemaker or implantable defibrillator, intracranial electrodes or other intracranial implant, abnormalities of the cranial vault opposite stimulation electrodes (plates, prostheses, uncovered skull)
* Recruitment in other interventional studies for the duration of the participation.
* Pregnant women and nursing mothers
* Non-affiliation to a social security scheme (excluding AME) or non-beneficiary of such a scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the immediate effect of a single tACS session on the static visual field size of patients with chronic phase HH | Immediately after the intervention
  To evaluate the immediate effect of a single tACS session, under two different conditions of tACS stimulation (right frontal stimulation (FEF, Frontal Eye Fields) and contralateral occipito-parietal stimulation to the lesion (V1-IPS, primary visual cortex and intraparietal sulcus or intra-parietal furrow) on the static visual field size of patients with chronic phase HH

CONTACTS AND LOCATIONS:
Locations (1):
- GH Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sahraie A. Induced visual sensitivity changes in chronic hemianopia. Curr Opin Neurol. 2007 Dec;20(6):661-6. doi: 10.1097/WCO.0b013e3282f1c70f. PMID 17992086
- [Background] Schuett S, Dauner R, Zihl J. Line bisection in unilateral homonymous visual field defects. Cortex. 2011 Jan;47(1):47-52. doi: 10.1016/j.cortex.2010.01.008. Epub 2010 Jan 28. PMID 20172510
- [Background] Sergeeva EG, Henrich-Noack P, Bola M, Sabel BA. Brain-state-dependent non-invasive brain stimulation and functional priming: a hypothesis. Front Hum Neurosci. 2014 Nov 5;8:899. doi: 10.3389/fnhum.2014.00899. eCollection 2014. No abstract available. PMID 25414662
- [Background] Sabel BA, Fedorov AB, Naue N, Borrmann A, Herrmann C, Gall C. Non-invasive alternating current stimulation improves vision in optic neuropathy. Restor Neurol Neurosci. 2011;29(6):493-505. doi: 10.3233/RNN-2011-0624. PMID 22124039
- [Background] Zaehle T, Rach S, Herrmann CS. Transcranial alternating current stimulation enhances individual alpha activity in human EEG. PLoS One. 2010 Nov 1;5(11):e13766. doi: 10.1371/journal.pone.0013766. PMID 21072168
- [Background] Helfrich RF, Knepper H, Nolte G, Struber D, Rach S, Herrmann CS, Schneider TR, Engel AK. Selective modulation of interhemispheric functional connectivity by HD-tACS shapes perception. PLoS Biol. 2014 Dec 30;12(12):e1002031. doi: 10.1371/journal.pbio.1002031. eCollection 2014 Dec. PMID 25549264
- [Background] Alekseichuk I, Diers K, Paulus W, Antal A. Transcranial electrical stimulation of the occipital cortex during visual perception modifies the magnitude of BOLD activity: A combined tES-fMRI approach. Neuroimage. 2016 Oct 15;140:110-7. doi: 10.1016/j.neuroimage.2015.11.034. Epub 2015 Nov 23. PMID 26608246